CLINICAL TRIAL: NCT00979121
Title: Randomized Trial of Rosuvastatin for Acutely Injured Lungs From Sepsis
Brief Title: Statins for Acutely Injured Lungs From Sepsis
Acronym: SAILS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: stopped for futility
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 670; N01HR056179 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2014-08

CONDITIONS: Sepsis; Acute Lung Injury
Keywords: ALI; Sepsis; statin
MeSH Terms: conditions — Sepsis; Acute Lung Injury | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): Half of the subjects were randomized to the active drug (Rosuvastatin).
  Dosage, Form, and Frequency: drug was provided as 10mg tablets and administered through an enteral feeding tube or orally (following extubation when patients were able to safely take oral medications). An initial 40mg loading dose was administered followed by a daily 20 mg maintenance dose. Maintenance dosing was adjusted for renal failure not compensated by renal replacement therapy.
  Duration: drug was administered daily until:
  1. 28 days after randomization or 3 days after ICU discharge (whichever comes first),
  2. Discharge from study hospital,
  3. Death
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Half of the subjects were randomized to placebo.
  10mg tablets identical to active drug were administered through an enteral feeding tube or orally (following extubation when patients were able to safely take oral medications). Dosage, frequency, and duration was provided in the same manner as the active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Subjects received an initial 40mg loading dose followed by 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharged from the study hospital.
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — Subjects received placebo by mouth or feeding tube daily for 28 days or until discharged from study hospital.
  Arms: Placebo

SUMMARY:
Objective: assess the efficacy and safety of oral rosuvastatin in patients with sepsis-induced Acute Lung Injury (ALI).

Hypothesis: Rosuvastatin therapy will improve mortality in patients with sepsis-induced ALI.

DETAILED DESCRIPTION:
Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS) involves extensive inflammation in the lungs that can lead to rapid respiratory failure. These conditions are most commonly caused by pneumonia, generalized infection, or severe trauma to the lungs, but can also be less commonly caused by smoke or salt water inhalation, drug overdose, or shock.

For some people, ALI/ARDS resolves without treatment, but many severe cases result in hospitalization in the intensive care unit (ICU), where 30% to 40% of cases end in mortality. Current treatments for ALI/ARDS include assisted breathing with a ventilator, supportive care, and management of the underlying causes.

Upon admission to the ICU, Rosuvastatin or placebo was administered through an enteral feeding tube or administered orally following extubation when patients were able to safely take oral medications. The type and placement of the enteral feeding tube (nasogastric, nasoenteric, PEG, orogastric, oroenteric, etc.) and the ability to safely take oral medications was determined by the patient's primary team. Study drug was blinded with an identical appearing placebo. The first study drug dose (rosuvastatin or placebo) was administered within 4 hours of randomization as a loading dose of 40 mg.

Blood pressure, heart rate, ventilation settings, and various blood factors were measured during treatment. Phone-based follow-up assessments occurred at months 6 and 12 after ICU discharge and included measurements of health-related quality of life; psychological, neurocognitive, and physical activity outcomes; healthcare utilization; and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1. Systemic inflammatory response syndrome (SIRS) defined as meeting at least criteria (a) or (b)for a systemic inflammatory response:

  1. White blood cell count >12,000 or <4,000 or >10% band forms
  2. Body temperature >38 degrees Celsius (C) (any route) or <36 degrees C (accepting core temperatures only; indwelling catheter, esophageal, rectal)
  3. Heart rate (> 90 beats/min) or receiving medications that slow heart rate or paced rhythm 2. Suspected or proven infection: Sites of infection include thorax, urinary tract, abdomen, skin, sinuses, central venous catheters, and bacterial meningitis (Appendix A).

     3. ALI as defined by acute onset of:

  <!-- -->

  1. PaO2 / FiO2 ≤ 300 (intubated). If altitude > 1000m, then PaO2 / FiO2 ≤ 300 x (PB/760), and
  2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph, and
  3. Requirement for positive pressure ventilation via an endotracheal tube, and
  4. No clinical evidence of left atrial hypertension, or if measured, a Pulmonary Arterial Wedge Pressure (PAOP) less than or equal to 18 mm Hg. If a patient has a PAOP > 18 mmHg, then the other criteria must persist for more than 12 hours after the PAOP has declined to ≤ 18 mmHg, and still be within the 48-hour enrollment window.

"Acute onset" is defined as follows: the duration of the hypoxemia criterion (#1) and the chest radiograph criterion (#2) must be ≤ 28 days at the time of randomization. Opacities considered "consistent with pulmonary edema" include any patchy or diffuse opacities not fully explained by mass, atelectasis, or effusion or opacities known to be chronic (> 28 days). The findings of vascular redistribution, indistinct vessels, and indistinct cardiac borders are not considered "consistent with pulmonary edema".

All ALI criteria (3a-d above) must occur within the same 24 hour period. The onset of ALI is when the last ALI criterion is met. Patients must be enrolled within 48 hours of ALI onset and no more than 7 days from the initiation of mechanical ventilation. SIRS criteria must occur within the 72 hours before or the 24 hours after ALI onset. Information for determining when these time window criteria were met may come from either the Network hospital or a referring hospital reports.

Exclusion Criteria:

1. No consent/inability to obtain consent
2. Age less than 18 years
3. More than 7 days since initiation of mechanical ventilation
4. More than 48 hours since meeting ALI inclusion criteria
5. Patient, surrogate, or physician not committed to full support ).
6. Unable to receive or unlikely to absorb enteral study drug
7. Rosuvastatin specific exclusions

   * Receiving a statin medication within 48 hours of randomization
   * Allergy or intolerance to statins
   * Physician insistence for the use or avoidance of statins during the current hospitalization
   * Creatine Kinase (CK) , alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal
   * Diagnosis of hypothyroidism and not on thyroid replacement therapy
   * Pregnancy or breast feeding
   * Receiving niacin, fenofibrate or cyclosporine, gemfibrozil, atazanavir, lopinavir, ritonavir, daptomycin
8. Severe chronic liver disease
9. Moribund patient not expected to survive 24 hours
10. Chronic respiratory failure defined as PaCO2 > 60 mm Hg in the outpatient setting
11. Home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for CPAP/BIPAP (Continuous Positive Airway Pressure/BiLevel Positive Airway Pressure) used solely for sleep-disordered breathing
12. Diffuse alveolar hemorrhage from vasculitis
13. Burns > 40% total body surface
14. Interstitial lung disease of severity sufficient to require continuous home oxygen therapy
15. Unwillingness or inability to utilize the ARDS network 6 ml/kg Predicted Body Weight (PBW) ventilation protocol
16. Cardiac disease classified as NYHA (New York Heart Association) class IV
17. Myocardial infarction within past 6 months
18. Intraparenchymal Central Nervous System (CNS) bleed within a month of randomization.
19. Temperature >40.3 C in the 6 hours before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Truwit, MD, Study Chair — University of Virginia, Medical Center
Locations (40):
- United States (40):
  - University of San Francisco-Fresno Medical Center, Fresno, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSF-Moffitt Hospital, San Francisco, California
  - University of California, San Francisco (UCSF)-Moffitt Hospital, San Francisco, California
  - Centura St. Anthony Central Hospital, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baton Rouge General Hospital-Blue Bonnet, Baton Rouge, Louisiana
  - Baton Rouge General Hospital-Midcity, Baton Rouge, Louisiana
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Medical Center of Louisiana, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland Shock Trauma Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Rochester Methodist Hospital, Rochester, Minnesota
  - St. Mary's Hospital, Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Durham Regional Medical Center, Durham, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - Wesley Long Community Hospital, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Providence Hospital, Everett, Washington
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Yu SY, Ge ZZ, Xiang J, Gao YX, Lu X, Walline JH, Qin MB, Zhu HD, Li Y. Is rosuvastatin protective against sepsis-associated encephalopathy? A secondary analysis of the SAILS trial. World J Emerg Med. 2022;13(5):367-372. doi: 10.5847/wjem.j.1920-8642.2022.072. PMID 36119770
- [Derived] Dinglas VD, Hopkins RO, Wozniak AW, Hough CL, Morris PE, Jackson JC, Mendez-Tellez PA, Bienvenu OJ, Ely EW, Colantuoni E, Needham DM. One-year outcomes of rosuvastatin versus placebo in sepsis-associated acute respiratory distress syndrome: prospective follow-up of SAILS randomised trial. Thorax. 2016 May;71(5):401-10. doi: 10.1136/thoraxjnl-2015-208017. Epub 2016 Mar 2. PMID 26936876
- [Derived] Needham DM, Colantuoni E, Dinglas VD, Hough CL, Wozniak AW, Jackson JC, Morris PE, Mendez-Tellez PA, Ely EW, Hopkins RO. Rosuvastatin versus placebo for delirium in intensive care and subsequent cognitive impairment in patients with sepsis-associated acute respiratory distress syndrome: an ancillary study to a randomised controlled trial. Lancet Respir Med. 2016 Mar;4(3):203-12. doi: 10.1016/S2213-2600(16)00005-9. Epub 2016 Jan 29. PMID 26832963
- [Derived] National Heart, Lung, and Blood Institute ARDS Clinical Trials Network; Truwit JD, Bernard GR, Steingrub J, Matthay MA, Liu KD, Albertson TE, Brower RG, Shanholtz C, Rock P, Douglas IS, deBoisblanc BP, Hough CL, Hite RD, Thompson BT. Rosuvastatin for sepsis-associated acute respiratory distress syndrome. N Engl J Med. 2014 Jun 5;370(23):2191-200. doi: 10.1056/NEJMoa1401520. Epub 2014 May 18. PMID 24835849
- See also: ARDS Network Website — http://www.ardsnet.org
- Available data/document: Individual Participant Data Set: ARDSNet-SAILS — http://biolincc.nhlbi.nih.gov/studies/sails/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/sails/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/sails/

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosuvastatin: Half of the subjects will receive the active drug, Rosuvastatin.
  Rosuvastatin: Patients will receive 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharged from the study hospital.
- Placebo: Half of the patients will be randomized to the placebo.
  Placebo: Patients will receive one placebo by mouth or feeding tube daily for 28 days or until discharged form study hospital.
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo
Started | 379 | 366
Completed | 379 | 366
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo | Total
Number analyzed (Participants) | 379 | 366 | 745
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 262 | 272 | 534
  >=65 years | 114 | 92 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (17.1) | 54.1 (15.6) | 54.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 185 | 380
  Male | 184 | 181 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 40 | 86
  Not Hispanic or Latino | 333 | 326 | 659
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 52 | 53 | 105
  White | 289 | 301 | 590
  More than one race | NA — not captured | NA — not captured | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 379 | 366 | 745
APACHE III Score [Mean (Standard Deviation); unit: units on a scale] — APACHE III Score: Acute, Physiology, Age, Chronic Health Evaluation III Prognostic System is a measure of hospital mortality risk for critically ill adult patients. Our study used a refined version based on the study by Knause and colleagues (Chest, 1991; 100:1619-36). The score is based on results from addition of 3 groups of variables (physiology, range: 0-252; age: 0-23; and chronic health: 0-24). Overall score range: 0-299; higher number indicates higher risk.
  units on a scale | 92.1 (28.4) | 94.8 (27.9) | 93.4 (28.2)
Primary cause of lung injury [Number; unit: participants] — Based on coding of primary vs. secondary by the site; data entry errors account for total count discrepancy.
  participants
    Aspiration | 26 | 23 | 49
    Multiple Transfusion | 3 | 1 | 4
    Other | 7 | 4 | 11
    Pneumonia | 267 | 260 | 527
    Sepsis | 72 | 73 | 145
    Trauma | 2 | 4 | 6
Baseline Shock [Number; unit: participants] — The number of participants who were in shock at the time of randomization. Baseline shock was defined as meeting one of the following conditions: a mean arterial pressure less than 60 mm Hg, receiving a vasopressor (norepinephrine, epinephrine, vasopressin or neosynephrine) at any dose, or receiving dopamine at a dose greater than or equal to 6 mcg/kg/min (or mcg/min) .
  participants | 173 | 166 | 339
PaFiO2:FiO2 ratio less than or equal to 200 mm Hg [Number; unit: participants] — The number of participants with a P/F ratio of 200 mm Hg or less at baseline.
  participants | 267 | 253 | 520
Hours from intubation to randomization [Number; unit: participants]
  24 hours or less | 124 | 129 | 253
  between 24 and 48 hours | 204 | 192 | 396
  between 48 and 72 hours | 41 | 31 | 72
  more than 72 hours | 10 | 13 | 23
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality to Day 60.
Description: The percentage of subjects alive at study day 60. Those subjects discharged home prior to day 60 were counted as alive at day 60.
Time Frame: 60 days after randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rosuvastatin: Half of the subjects were randomized to active drug (Rosuvastatin).
  Rosuvastatin: Subjects received 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharge from the study hospital.
- Placebo: Half of the subjects were randomized to placebo.
  Placebo: Subjects received placebo by mouth or feeding tube daily for 28 days or until discharge from study hospital.
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 379 | 366
percentage of participants | 28.5 [24.0 to 33.0] | 24.9 [20.5 to 29.3]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Hospital mortality to day 60 was estimated using the Kaplan Meier estimate, with patients discharged home before day 60 considered alive at day 60. The analysis was stratified by co-enrolled treatment assignments for 81 patients also enrolled in a randomized clinical trial of two different nutritional strategies. A maximum of 1000 patients were to be enrolled, providing a 92% probability of rejecting the null hypothesis for the effect on mortality if a true difference in mortality was 9%; Test type: Superiority or Other; p = 0.21, Proc lifetest — The monitoring boundaries were designed to have a low probability of stopping for futility before 750 patients. The maximum sample size was 1000 patients. Efficacy stopping was based on mortality; futility stopping was based on mortality and VFDs; Proc lifetest was used to calculate mortality mean and variance due to one subject lost to follow up who was censored; difference in % of pts alive at 60 days = 4.0, 95% CI 2-sided [-2.3 to 10.2]

2. Secondary Outcome: Ventilator Free Days at Study Day 28
Description: Ventilator Free Days (VFDs) to day 28 were defined as the number of days from the time of initiating unassisted breathing to day 28 after randomization, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a subject received assisted breathing at day 27 or died prior to day 28, a value of zero VFDs was given.
Time Frame: time of initiating unassisted breathing to day 28 after study randomization
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo: Half of the subjects were randomized to placebo.
  Placebo: Subjects received placebo by mouth or feeding tube daily for 28 days or until discharged from study hospital.
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 379 | 366
days | 15.1 (10.8) | 15.1 (11.0)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Ventilator, ICU free, and organ failure free days were analyzed by analysis of variance, utilizing treatment assignment where applicable; Test type: Superiority or Other; p = 0.96, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI [-1.6 to 1.5]

3. Other Pre Specified Outcome: Organ Failure Free Days at Day 14
Description: The number of days from randomization to day 14 without an organ failure. Four main organ systems were measured: cardiovascular, coagulation, hepatic function, and renal function.
Time Frame: 14 days after randomization
Measure: Mean (Standard Deviation); unit: days
Groups:
- Rosuvastatin: Half of the subjects were randomized to active drug (Rosuvastatin).
  Rosuvastatin: Patients received 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharge from the study hospital.
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 379 | 366
days
  Cardiovascular | 8.5 (4.8) | 8.7 (4.9)
  Coagulation | 10.7 (5.1) | 11.1 (4.8)
  Hepatic | 10.8 (5.0) | 11.8 (4.3)
  Renal | 10.1 (5.3) | 11.0 (4.7)

4. Other Pre Specified Outcome: ICU Free Days to Day 28
Time Frame: 28 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 379 | 366
days | 14.3 (10.1) | 14.4 (10.3)

5. Other Pre Specified Outcome: Other Secondary Out-comes
Description: Percentage of subjects with Arrhythmia's, Bowel Ischemia, Myocardial Infarction, Ischemic Stroke, and Thromboembolism were measured.
Time Frame: 28 days after randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 367 | 360
percentage of participants
  Arrhythmias | 9.0 [6.1 to 11.9] | 8.4 [5.5 to 11.3]
  Bowel Ischemia | 1.4 [0.2 to 2.6] | 1.9 [0.5 to 3.3]
  Myocardial Infarction | 0.5 [-0.3 to 1.3] | 0.6 [-0.2 to 1.4]
  Ischemic Stroke | 0.3 [-.03 to 0.9] | 0.3 [-0.3 to 0.9]
  Thromboembolism | 6.3 [3.8 to 8.9] | 6.9 [4.4 to 9.5]

6. Other Pre Specified Outcome: Changes in Plasma Concentrations of C-reactive Protein (CRP) From Baseline to Day 6 and Day 14
Description: CRP levels were collected on subjects at baseline and on-study. The change in concentration from baseline levels to levels on study days 6 and 14 was analyzed. Those subjects that were still alive and on study at day 6 and 14 with a measured CRP level were included in the analysis.
Time Frame: 6 and 14 days after randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Rosuvastatin: Half of the subjects were randomized to active drug (Rosuvastatin).
  Rosuvastatin:Subjects received 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharge from the study hospital.
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 229 | 229
mg/dL
  Day 6 | -12.9 (27.79) | -15.1 (23.26)
  Day 14 | -19.8 (31.23) | -14.8 (26.28)

ADVERSE EVENTS:
Time Frame: Investigators conducted daily assessments for the presence of adverse events (AE) from enrollment through study day 28 or hospital discharge, whichever occurred first.
Description: AE definition: any clinically important untoward medical occurrence in a patient receiving study drug/procedures which was different than expected in the clinical course of a patient with ALI or an occurrence thought to be associated with the study drug/procedures. CK, ALT/AST at specified levels and CNS bleed were also systematically reported.
Groups:
- Rosuvastatin: Half of the subjects were randomized to the active drug (Rosuvastatin).
  Rosuvastatin: Subjects received 20 mg of study drug daily by mouth or feeding tube for 28 days or until discharge from the study hospital.
Arm/Group | Rosuvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 34/379 | 32/366
Other Adverse Events (participants affected / at risk) | 0/379 | 0/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=379) | Placebo (N=366)
Hemorrhage Retroperitoneal (General disorders) | 1 (1) | 1 (1)
Hyperpyrexia (General disorders) | 2 (2) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Neuroleptic Malignant Syndrome (General disorders) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 3 (3) | 4 (4)
Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hemorrhage (Nos) (Cardiac disorders) | 1 (1) | 0 (0)
Thrombosis Venous Arm (Cardiac disorders) | 1 (1) | 0 (0)
Venous Thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
ALT > 8 times upper limit of normal (Gastrointestinal disorders) | 0 (0) | 3 (3)
Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischemia Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrosis Bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction Small Intestine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peforation Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
AST > 8 times upper limit of normal (Investigations) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Ast Increased (Investigations) | 1 (1) | 0 (0)
Creatinine Serum Increased (Investigations) | 0 (0) | 1 (1)
CK > 10 times upper limit of normal (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Brain Disorder (Nos) (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracerebral Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Coughing Blood (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Failure Kidney Acute (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
sponsor can review results communications prior to public release and can embargo communications regarding trial results until presented at the American Thoracic Society international meeting.